CLINICAL TRIAL: NCT04339699
Title: STITCH - Prospective Multi Center Comparative Parallel Concurrent Study of the NobleStitch EL Compared to FDA Approved Amplatzer Occluder Device for Closure of Patent Foramen Ovale to Prevent Recurrent Ischemic Stroke
Brief Title: NobleStitch EL STITCH Trial is a PFO Comparative Trial
Acronym: STITCH
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor has voluntarily suspended Trial, to update Protocol and respond to observations by the FDA
Sponsor: Nobles Medical Technologies II Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 748824-0819; NCT05025475 (obsolete NCT alias)
Record Dates: First submitted 2020-04-01; First posted 2020-04-09 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Foramen Ovale, Patent; Stroke, Ischemic
Keywords: Patent Foramen Ovale; Stroke
MeSH Terms: conditions — Foramen Ovale, Patent; Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: A 640 participants indicated for percutaneous transcatheter closure of a PFO to reduce risk of recurrent Ischemic Stroke; between ages 18 - 60 years, who have had a Cryptogenic Stroke due to Paradoxical Embolism. To be conducted both in the USA and the European Union.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- NobleStitch™EL (Active Comparator): Participants treated with the NobleStitch™EL device
  Interventions: Device: NobleStitch™EL Suture Mediated Closure System
- Amplatzer PFO Occluder (Active Comparator): Participants treated with the Amplatzer PFO Occluder device
  Interventions: Device: Amplatzer PFO Occluder

INTERVENTIONS:
Device: NobleStitch™EL Suture Mediated Closure System — Percutaneous closure of Patent Foramen Ovale (PFO) using NobleStitch™EL suture Medicate Closure System
  Arms: NobleStitch™EL
Device: Amplatzer PFO Occluder — Percutaneous closure of Patent Foramen Ovale (PFO) using Amplatzer PFO Occluder
  Arms: Amplatzer PFO Occluder

SUMMARY:
STITCH - Prospective Multi-Center Comparative Parallel Concurrent Study of the NobleStitch™ EL versus FDA-approved Amplatzer Occluder device for closure of Patent Foramen Ovale to prevent recurrent Ischemic stroke.

DETAILED DESCRIPTION:
To demonstrate the non-inferiority of the NobleStitch™ EL with medical management in both safety and effectiveness compared to the FDA-approved Amplatzer Occluder with medical management for PFO Closure.

To demonstrate that the NobleStitch EL does not increase the incidence of ischemic stroke compared to published medical management data.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female ages 18 - 60 years old
* A PFO and a Cryptogenic Stroke verified by a neurologist
* Stroke is defined as an acute focal neurological deficit, presumed to be due to focal ischemia, and either:

  * Symptoms persisting ≥24 hours, or
  * Symptoms persisting <24 hours with Magnetic Resonance or CT findings of a new, neuroanatomical relevant infarct
* Cryptogenic stroke was defined as a stroke of unknown cause
* Prolonged cardiac rhythm monitoring (recommended 30 days and not less than 24 hours required)
* Intra and extracranial artery imaging: Magnetic Resonance Angiography, CT angiography, or contrast angiography, or contrast angiography or echocardiography of the carotid arteries to rule out ischemic stroke associated with atherosclerotic plaque, arterial dissection, or other vascular diseases. (The aortic arch may also be evaluated by TEE).
* Hypercoagulable state assessment to rule out an underlying hypercoagulable state

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning a pregnancy during the course of the study
* Age <18 or > 60 years of age
* Previous myocardial infarction or unstable angina within 6 months
* Clinically significant mitral or aortic valve stenosis or severe regurgitation
* Left Ventricular Ejection Fraction <50 percent
* Progressive neurological dysfunction or reduced life expectancy
* Contrast allergy
* Atrial Septal Defect (baseline left to right shunt assessed by TEE or other congenital heart diseases
* Active Endocarditis
* Perspective participants with known causes of Ischemic Stroke
* Arterial dissection
* Contraindicated or unsuitable for antiplatelet agents or oral anticoagulants
* Perspective participants with prosthetic heart valves
* Uncontrolled diabetes Mellitus
* Pulmonary hypertension
* Uncontrolled systemic hypertension
* Intracranial pathology
* Neurological deficits not due to stroke that may affect neurologic assessments
* Active autoimmune disease
* Active infection
* Alcohol and/or drug abuse
* A requirement for chronic anticoagulation therapy that cannot be discontinued
* Anatomic features (inability to achieve vascular access)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 640 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Effective PFO closure rate of the NobleStitch EL | 6 months
  Effectiveness PFO closure rate of NobleStitch EL suture mediated closure with medical management compared to Amplatzer PFO occluder with medical management for PFO closure. Effective PFO closure rate defined as Grade 0 or 1 shunt at rest and during Valsalva at 6 month post closure attempts

SECONDARY OUTCOMES:
Decreased event rate of recurrent ischemic stroke following PFO closure using NobleStitch EL | 5 years
  Safety of NobleStitch EL suture mediated closure system as compared to Amplatzer PFO Occluder Procedural and device related adverse event rate at 6 month follow up recurrent ischemic stroke through 5 years follow up

OTHER OUTCOMES:
The occurrence of recurrent ischemic stroke post procedural of patent foramen ovale closure | 5 Years
  Examination of Recurrent Ischemic Stroke through 5 year follow up. Comparison of the rate of Stroke associated with the NobleStitch EL procedure to that expected with medical management

CONTACTS AND LOCATIONS:
Overall Officials: Anthony A Nobles, PhD, Study Director — Nobles Medical Technologies II Inc
Locations (5):
- United States (4):
  - TMC HealthCare, Tucson, Arizona
  - USF/Tampa General Hospital, Tampa, Florida
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Inova Structural Heart Disease Program - Fairfax, Fairfax, Virginia
- Ospedale S. Eugenio, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) from the completed STITCH clinical trial that underlie the results reported in the Study, shall after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Immediately the following publication and ending 24 months after publication
Access Criteria: Will be available to Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. It will be available for Individual participant data meta-analysis

REFERENCES:
- [Background] Gaspardone A, De Marco F, Sgueglia GA, De Santis A, Iamele M, D'Ascoli E, Tusa M, Corciu A, Mullen M, Nobles A, Carminati M, Bedogni F. Novel percutaneous suture-mediated patent foramen ovale closure technique: early results of the NobleStitch EL Italian Registry. EuroIntervention. 2018 Jun 8;14(3):e272-e279. doi: 10.4244/EIJ-D-18-00023. PMID 29616629